CLINICAL TRIAL: NCT02782559
Title: Randomized Double-Blind, Placebo Controlled Evaluation of the Efficacy of Sildenafil Versus Placebo in Preterm Preeclampsia
Brief Title: Efficacy of Sildenafil in Preterm Preeclampsia
Acronym: SIL
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: difficulties acquiring the drug and funding for the drug
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-16-0083
Record Dates: First submitted 2016-02-11; First posted 2016-05-25 (Estimated); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Preterm Preeclampsia
MeSH Terms: interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sildenafil (Experimental): Sildenafil 40mg oral tablet three times a day from randomization until delivery
  Interventions: Drug: Sildenafil
- Placebo (Placebo Comparator): Matched to oral capsule of active treatment three times a day from randomization until delivery
  Interventions: Drug: Sildenafil; Drug: Placebo

INTERVENTIONS:
Drug: Sildenafil
Drug: Placebo — Color and size matched to active drug (sildenafil)
  Arms: Placebo

SUMMARY:
Randomized controlled trial to assess efficacy of Sildenafil in addition to expectant management for the treatment of preterm preeclampsia

DETAILED DESCRIPTION:
Preeclampsia is a major cause of maternal mortality. When preeclampsia presents prior to thirty-four weeks of gestation, expectant management is the standard practice in stable patients with the goal of extending pregnancy and therefore decreasing the risk of adverse outcomes in the premature neonate. Our aim was to assess the efficacy of Sildenafil, a phosphodiesterase inhibitor, versus placebo, in addition to expectant management, for the treatment of preterm preeclampsia to prolong pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients of gestational age of ≥24 0/7 weeks to ≤32 0/7 weeks.
2. Dating of pregnancy by ultrasound < or equal to 22 weeks or IVF conception
3. Diagnosis of Preterm Preeclampsia or Superimposed Preeclampsia

Exclusion Criteria:

1. Need for immediate delivery of the fetus
2. Known lethal anomaly
3. Pre-existing renal disease
4. Hypersensitivity to sildenafil
5. Pre-gestational diabetes, class C (onset prior to 10-19 or duration 10-19 yrs
6. Active peptic ulcer disease
7. Undergoing nitrate therapy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Latency (duration of pregnancy from diagnosis/randomization until delivery) | Diagnosis (randomization) until delivery, up to 34 weeks)
  earliest randomization can occur at 24 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Robyn P Roberts, MD, Principal Investigator — The University of Texas Health Science Center, Houston

IPD SHARING:
Plan to Share IPD: Yes